CLINICAL TRIAL: NCT00589979
Title: Efficacy and Safety of the Lidocaine 5% Patch When Used as Adjunct Treatment in Patients With Osteoarthritis of the Knee Receiving Sub-Optimal Pain Relief From Their Current Analgesic Regimen
Brief Title: Efficacy and Safety of the Lidoderm Patch Applied to Patients With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: EN3260-003
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Results first posted 2010-09-22 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis; Knee; Lidoderm; Lidocaine; Topical patch; Adjunct therapy
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Lidoderm; Lidocaine; Transdermal Patch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidoderm (Lidocaine 5% Patch) (Experimental): Lidoderm (lidocaine 5% patch) 10cm X 14cm patches each on the front and back of the index knee every 24 hours (q24h)
  Interventions: Drug: Lidoderm (Lidocaine 5% Patch)
- Placebo Patch (Placebo Comparator): Placebo Patch 10cm X 14cm patches each on the front and back of the index knee every 24 hours (q24h)
  Interventions: Drug: Placebo Patch

INTERVENTIONS:
Drug: Lidoderm (Lidocaine 5% Patch) — Topical Patch
  Other Names: Lidoderm
  Arms: Lidoderm (Lidocaine 5% Patch)
Drug: Placebo Patch — Topical Patch
  Other Names: Placebo
  Arms: Placebo Patch

SUMMARY:
Patients with knee pain due to Osteoarthritis (OA) experiencing sub-optimal pain relief from their current analgesic regimen will participate in a pilot clinical trial to evaluate the effectiveness and tolerability of the Lidoderm Patch compared with placebo in treating knee pain from OA.

ELIGIBILITY:
Key Inclusion criteria:

* Male or female patients ≥37 years with moderate-to-severe OA related pain in one knee
* Body mass index (BMI) ≤40 kg/m2
* Symptomatic OA of the index knee diagnosed with a functional capacity of II or III according to ACR criteria classification Note: Patients with symptomatic contralateral knee OA with persistent pain ≤2 cm on a 0-10 cm PI-NRS for ≥2 months will be allowed to participate.
* Unchanged dose of analgesic medication for OA for at least 4 weeks prior to screening and for the duration of the study
* Able and willing to complete all paper and e-diary assessments required by protocol

Key Exclusion criteria:

* Pain in any joint other than the index joint that could interfere with the patient's assessment of pain in the index joint
* Compromised integrity of the intact, superficial skin layer
* A grade 1 or 4 Kellgren and Lawrence score on radiographic examination
* Recent injury to either knee causing pain and interference with daily activities (eg. walking)
* Recent surgery/procedure to either knee causing pain that could interfere with study assessments of pain, function, and QoL
* Known hypersensitivity or allergy to lidocaine, local anesthetics of the amide type, or any component of the product

Min Age: 37 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2007-03; Primary Completion 2008-06 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ernest A. Kopecky, PhD, MBA, Study Director — Endo Pharmaceuticals
Locations (20):
- United States (20):
  - Arizona Arthritis Research, PLC, Paradise Valley, Arizona
  - NextCare Institute for Clinical Research, Phoenix, Arizona
  - HOPE Research Institute, LLC, Phoenix, Arizona
  - Clinical Research Consulting, Milford, Connecticut
  - New England Research Associates, LLC, Trumbull, Connecticut
  - Tampa Bay Medical Research, Inc., Clearwater, Florida
  - Delray Research Associates, Delray Beach, Florida
  - CNS Clinical Trials, St. Petersburg, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Arthritis & Osteoporosis Center of Maryland, Frederick, Maryland
  - Midwest Pharmaceutical Research, City of Saint Peters, Missouri
  - Arthritis Center of Nebraska, Lincoln, Nebraska
  - Comprehensive Clinical Research, Berlin, New Jersey
  - University Hospitals of Case Medical Center - Arthritis Translational Research Program, Beachwood, Ohio
  - Community Research, Cincinnati, Ohio
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Health Concepts, Rapid City, South Dakota
  - Radiant Research, San Antonio, Texas
  - Advanced Pain Management & Rehabilitation, Hilltop Medical, Virginia Beach, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This exploratory, Phase IIb study was initiated on March 6, 2007 at 21 study centers in the United States and completed on June 24, 2008.
Pre-assignment Details: During the active Run-in Period, eligible patients applied Lidoderm patches every 24 hours for 28 days. During the 12-week Double-blind Treatment Period, patients were randomized to apply Lidoderm patches or matching placebo patches every 24 hours for 4 weeks and then crossed over to the other treatment for the next two 4-week treatment periods.
Groups:
- Run-in Period: Lidoderm: Run-in Period with patients applying Lidoderm (lidocaine 5% patch) 10cm x 14cm each on the front and back of the index knee every 24 hours for up to 28 days (4 weeks).
- Treatment Sequence: Lidoderm - Placebo - Placebo: Lidoderm (lidocaine 5% patch) 10cm X 14cm patches each on the front and back of the index knee every 24 hours (q24h) for up to 4 weeks followed by matching placebo 10cm x 14cm patches each on the front and back of the index knee q24h for up to 8 weeks
- Treatment Sequence: Placebo - Lidoderm - Lidoderm: Matching placebo 10cm X 14cm patches each on the front and back of the index knee q24h for up to 4 weeks followed by Lidoderm (lidocaine 5% patch) 10cm x 14cm patches each on the front and back of the index knee q24h for up to 8 weeks
Period: Run-In Period
Arm/Group | Run-in Period: Lidoderm | Treatment Sequence: Lidoderm - Placebo - Placebo | Treatment Sequence: Placebo - Lidoderm - Lidoderm
Started | 169 | 0 | 0
Completed | 93 | 0 | 0
Not Completed | 76 | 0 | 0
Not completed — Adverse Event | 5 | 0 | 0
Not completed — Protocol Violation | 3 | 0 | 0
Not completed — Did not qualify for randomization | 54 | 0 | 0
Not completed — Withdrawal by Subject | 10 | 0 | 0
Not completed — Informed Consent Withdrawn | 4 | 0 | 0
Period: Double-Blind Treatment Period 1
Arm/Group | Run-in Period: Lidoderm | Treatment Sequence: Lidoderm - Placebo - Placebo | Treatment Sequence: Placebo - Lidoderm - Lidoderm
Started | 0 (Participants completing the Run-in Period were then randomized to two different treatment sequences.) | 50 (N=21 randomized on or after 22JAN2008; included in mod. intent-to-treat (MITT) analysis population.) | 43 (N=21 randomized on or after 22JAN2008; included in mod. intent-to-treat (MITT) analysis population.)
Completed | 0 | 48 | 41
Not Completed | 0 | 2 | 2
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Period: Double-Blind Treatment Period 2
Arm/Group | Run-in Period: Lidoderm | Treatment Sequence: Lidoderm - Placebo - Placebo | Treatment Sequence: Placebo - Lidoderm - Lidoderm
Started | 0 | 48 (N=19 randomized on or after 22JAN2008; included in mod. intent-to-treat (MITT) analysis population.) | 41 (N=20 randomized on or after 22JAN2008; included in mod. intent-to-treat (MITT) analysis population.)
Completed | 0 | 47 | 39
Not Completed | 0 | 1 | 2
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Other | 0 | 0 | 1
Period: Double-Blind Treatment Period 3
Arm/Group | Run-in Period: Lidoderm | Treatment Sequence: Lidoderm - Placebo - Placebo | Treatment Sequence: Placebo - Lidoderm - Lidoderm
Started | 0 | 47 (N=19 randomized on or after 22JAN2008; included in mod. intent-to-treat (MITT) analysis population.) | 39 (N=19 randomized on or after 22JAN2008; included in mod. intent-to-treat (MITT) analysis population.)
Completed | 0 | 46 | 38
Not Completed | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Sequence: Lidoderm - Placebo - Placebo: Lidoderm (lidocaine 5% patch) 10cm X 14cm patches each on the front and back of the index knee every 24 hours (q24h) for 4 weeks followed by matching placebo 10cm x 14cm patches each on the front and back of the index knee q24h for up to 8 weeks.
- Sequence: Placebo - Lidoderm - Lidoderm: Matching placebo 10cm X 14cm patches each on the front and back of the index knee q24h for 4 weeks followed by Lidoderm (lidocaine 5% patch) 10cm x 14cm patches each on the front and back of the index knee q24h for up to 8 weeks.
- Total: Total of all reporting groups
Arm/Group | Sequence: Lidoderm - Placebo - Placebo | Sequence: Placebo - Lidoderm - Lidoderm | Total
Number analyzed (Participants) | 50 | 43 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (10.0) | 61.1 (10.9) | 61.1 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 28 | 60
  Male | 18 | 15 | 33
Region of Enrollment [Number; unit: participants]
  United States | 50 | 43 | 93

OUTCOME MEASURES:

1. Primary Outcome: Time-to-Exit From Current Study Treatment
Description: Time-to-exit was defined as the number of days at which a patient either met the switching criterion [a 2-category change in the Pain Relief Scale (PRS) score in the worsening direction (increasing pain or decreasing pain relief) for 2 consecutive days] or discontinued from the study. The PRS is a 9-point categorical rating scale to assess pain relief in the last 24 hours in which 0 = completely worse and 8 = complete pain relief. Traditional survival models that consider event times (e.g. median survival time) as independent and homogeneous across patients were not suitable for this study.
Time Frame: Baseline, Period 1 (up to 4 weeks ±2 days), Period 2 (up to 4 weeks ±2 days), Period 3 (up to 4 weeks ±2 days), or Premature Discontinuation
Population: The modified intent-to treat (MITT) population consisted of all intent-to-treat (ITT) patients who were randomized on or after January 22, 2008.
  Note: Kaplan-Meier estimates for median time-to-exit from current study treatment could not be calculated for Period 2 or Period 3, because the survival distribution function did not fall below 0.5000.
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- Sequence: Lidoderm - Placebo - Placebo (LPP): Lidoderm (lidocaine 5% patch) 10cm X 14cm patches each on the front and back of the index knee every 24 hours (q24h) for 4 weeks followed by matching 10cm x 14cm patches each on the front and back of the index knee q24h for up to 8 weeks
- Sequence: Placebo - Lidoderm - Lidoderm (PLL): Matching placebo 10cm X 14cm patches each on the front and back of the index knee every 24 hours (q24h) for 4 weeks followed by Lidoderm (lidocaine 5% patch) 10cm x 14cm patches each on the front and back of the index knee q24h for up to 8 weeks
Arm/Group | Sequence: Lidoderm - Placebo - Placebo (LPP) | Sequence: Placebo - Lidoderm - Lidoderm (PLL)
Number analyzed (Participants) | 21 | 21
Days
  Period 1 ( Sequence LPP, N=21; Sequence PLL, N=21) | 31 [10 to 31] | 20 [12 to 30]
  Period 2 (Sequence LPP, N=19; Sequence PLL, N=20) | NA [NA to NA] — Survival distribution function did not reach 0.5000; ie, patients within the study period did not reach exit criteria by the end of the 4-week period. | NA [NA to NA] — Survival distribution function did not reach 0.5000; ie, patients within the study period did not reach exit criteria by the end of the 4-week period.
  Period 3 (Sequence LPP, N=19; Sequence PLL, N=19) | NA [19 to NA] — Survival distribution function did not reach 0.5000; ie, patients within the study period did not reach exit criteria by the end of the 4-week period. | NA [NA to NA] — Survival distribution function did not reach 0.5000; ie, patients within the study period did not reach exit criteria by the end of the 4-week period.
Statistical Analysis 1: Comparison: Sequence: Lidoderm - Placebo - Placebo (LPP) vs Sequence: Placebo - Lidoderm - Lidoderm (PLL); The two treatments were compared by time-varying relative hazards, associated P values, and 95% confidence intervals. Appropriate survival or hazard functions were calculated; Test type: Superiority or Other; p = 0.1006, Cox frailty model — All statistical tests were 2-sided with a significance level of alpha=0.05; Model included treatment, sequence, period, and first-order carryover as fixed effects and frailty; patient nested within sequence was frailty; Hazard Ratio (HR) = 1.78, 95% CI [0.89 to 3.55] — The Hazard Ratio (HR) provided is the ratio of Placebo to Lidoderm

2. Secondary Outcome: Time-to-Exit Due to Lack of Efficacy
Description: Time-to-exit due to lack of efficacy was defined as a patient that met the switching criterion (a 2-category change in Pain Relief Scale (PRS) in the worsening direction [increasing pain or decreasing pain relief] for 2 consecutive days) or was discontinued from the current period or study due to lack of efficacy. The PRS is a 9-point categorical rating scale to assess pain relief in the last 24 hours in which 0 = completely worse and 8 = complete pain relief.
  No patients discontinued from the study due to lack of efficacy.
Time Frame: Period 1 (up to 4 weeks), Period 2 (up to 4 weeks), Period 3 (up to 4 weeks), or Premature Discontinuation
Population: The modified intent-to treat (MITT) population consisted of all intent-to-treat (ITT) patients who were randomized on or after January 22, 2008.
  Note: No patients exited a study period due to lack of efficacy, therefore median time-to-exit could not be calculated.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sequence: Lidoderm - Placebo - Placebo (LPP) | Sequence: Placebo - Lidoderm - Lidoderm (PLL)
Number analyzed (Participants) | 21 | 21
days
  Period 1 (Sequence LPP, N=21; Sequence PLL, N=21) | NA [NA to NA] — No patients discontinued from this study period due to lack of efficacy. | NA [NA to NA] — No patients discontinued from this study period due to lack of efficacy.
  Period 2 (Sequence LPP, N=19; Sequence PLL, N=20) | NA [NA to NA] — No patients discontinued from this study period due to lack of efficacy. | NA [NA to NA] — No patients discontinued from this study period due to lack of efficacy.
  Period 3 (Sequence LPP, N=19; Sequence PLL, N=19) | NA [NA to NA] — No patients discontinued from this study period due to lack of efficacy. | NA [NA to NA] — No patients discontinued from this study period due to lack of efficacy.

3. Secondary Outcome: Exit Status From Current Study Treatment - Yes
Description: Exit status from a current study treatment was categorized as yes or no for patients who exited prior to the 4-week planned duration. This analysis supports the results of the primary analysis. The number of patients exiting (yes) is reported.
Time Frame: Baseline, Period 1 (up to 4 weeks), Period 2 (up to 4 weeks), Period 3 (up to 4 weeks), or Premature Discontinuation
Population: The modified intent-to-treat (MITT) population consisted of all intent-to-treat (ITT) patients defined as all patients who received study medication and provided run-in and baseline assessments and had at least 1 post-baseline efficacy assessment and who were randomized on or after January 22, 2008.
Measure: Number; unit: Participants
Arm/Group | Sequence: Lidoderm - Placebo - Placebo (LPP) | Sequence: Placebo - Lidoderm - Lidoderm (PLL)
Number analyzed (Participants) | 21 | 21
Participants
  Period 1 (Sequence LPP, N=21; Sequence PLL, N=21) | 10 | 12
  Period 2 (Sequence LPP, N=19; Sequence PLL, N=20) | 5 | 4
  Period 3 (Sequence LPP, N=19; Sequence PLL, N=19) | 6 | 2
Statistical Analysis 1: Comparison: Sequence: Lidoderm - Placebo - Placebo (LPP) vs Sequence: Placebo - Lidoderm - Lidoderm (PLL); The proportion of patients who exited from the current treatment period prior to the 4-week planned duration was analyzed using a logistic regression model for repeated measures; Test type: Superiority or Other; p = 0.1272, Regression, Logistic — The logistic regression model for repeated measures used for this analysis included treatment, sequence, period, and first-order carry-over as fixed effects and repeated measures taken on patients nested within sequence; The results presented are reported in terms of odds ratios, corresponding 95% confidence intervals, and P-values for each fixed effect in the model; Odds Ratio (OR) = 1.86, 95% CI [0.86 to 4.02] — The Odds Ratio (OR) provided is the ratio of Lidoderm to Placebo

4. Secondary Outcome: Overall Treatment Difference in the LSMeans of the Average of the Last Two Daily Pain Intensity Numerical Rating Scale (PI-NRS)
Description: The Numerical Rating Scale (NRS) is an 11-point categorical rating scale to assess pain intensity (PI-NRS); 0= no pain and 10= worst possible pain. The scale is anchored on the left with "No Pain" and on the right with "Worst Possible Pain." Patients were to complete this assessment at approximately the same time each day during the double-blind treatment period in their e-diary. The overall treatment difference for the Lidoderm (lidocaine patch 5%) and placebo patch was compared by combining data for patients receiving the respective treatment regardless of the randomized study sequence.
Time Frame: Baseline, End of Period 1 (up to 4 weeks), End of Period 2 (up to 4 weeks) and End of Period 3 (up to 4 weeks)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Lidoderm (Lidocaine 5% Patch): The group represents the pooled data for all patients receiving Lidoderm (lidocaine 5% patch) during the randomized, double-blind treatment period regardless of the randomized study sequence.
- Placebo Patch: The group represents the pooled data for all patients receiving Placebo patches during the randomized, double-blind treatment period regardless of the randomized study sequence.
Arm/Group | Lidoderm (Lidocaine 5% Patch) | Placebo Patch
Number analyzed (Participants) | 21 | 21
Units on a scale | 3.03 (0.35) | 3.57 (0.35)
Statistical Analysis 1: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; The overall treatment difference for the lidocaine patch 5% and placebo patch was compared by combining data for patients receiving the respective treatment regardless of the randomized study sequence. The endpoint was analyzed by linear mixed effects models incorporating treatment, period, sequence, and first-order carryover as fixed effects, and patient nested within sequence as a random effect. P-value for the random effect (s2) is from the Wald Z-test for the covariance parameter estimates; Test type: Superiority or Other; p = 0.0224, Linear mixed effects model — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = -0.54, 95% CI [-1.01 to -0.08] — The results are reported as least squares means and their differences along with associated P-values, and 95% confidence intervals for each fixed effect in the model

5. Secondary Outcome: Overall Treatment Difference in the LSMeans of the Average of the Last Two Daily Pain Relief Scale (PRS) Scores
Description: The Pain Relief Scale (PRS) is a 9-point categorical rating scale to assess pain relief during the 24-hours since the last assessment; 0= completely worse and 8= complete pain relief. Patients completed this assessment each day during the run-in period and each day during the double-blind treatment phase in their e-diary.
Time Frame: Baseline, End of Period 1 (up to 4 weeks), End of Period 2 (up to 4 weeks) and End of Period 3 (up to 4 weeks)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Lidoderm (Lidocaine 5% Patch) | Placebo Patch
Number analyzed (Participants) | 21 | 21
Units on a scale | 4.45 (0.25) | 4.06 (0.25)
Statistical Analysis 1: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.2747, Linear mixed effects regression — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = 0.39, 95% CI [-0.31 to 1.09] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Overall Treatment Difference of the LSMeans of the Pain Quality Assessment Scale (PQAS) Scores
Description: The PQAS measures individual pain qualities and the impact of treatment on those qualities. Items 1-19 are each rated on an 11-point scale ranging from 0 (lowest score - no pain of that type) to 10 (highest score - the highest level of that type of pain). Average surface pain = average of PQAS items: cold, sensitive, itchy, numb, and tingling. Average deep pain = average of PQAS items: dull, cramping, throbbing, aching, and heavy. Average paroxymal pain = average of PQAS items: sharp, shooting, electric, and radiating.
Time Frame: Baseline, Period 1 (up to 4 weeks), Period 2 (up to 4 weeks), Period 3 (up to 4 weeks)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Lidoderm (Lidocaine 5% Patch) | Placebo Patch
Number analyzed (Participants) | 21 | 21
Units on a scale
  Intense | 3.31 (0.32) | 3.53 (0.32)
  Sharp | 2.50 (0.34) | 3.00 (0.34)
  Hot | 1.12 (0.26) | 1.59 (0.27)
  Dull | 3.04 (0.33) | 3.28 (0.33)
  Cold | 0.62 (0.14) | 0.50 (0.14)
  Sensitive | 0.88 (0.20) | 0.96 (0.21)
  Tender | 2.08 (0.30) | 1.89 (0.30)
  Itchy | 0.90 (0.23) | 1.00 (0.23)
  Shocking | 1.95 (0.34) | 2.36 (0.34)
  Numb | 1.31 (0.28) | 1.52 (0.28)
  Electrical | 1.32 (0.29) | 1.26 (0.30)
  Tingling | 1.24 (0.26) | 1.24 (0.26)
  Cramping | 1.78 (0.33) | 2.03 (0.33)
  Radiating | 2.03 (0.35) | 2.10 (0.35)
  Throbbing | 2.24 (0.34) | 2.06 (0.35)
  Aching | 2.78 (0.36) | 3.22 (0.37)
  Heavy | 2.12 (0.34) | 2.26 (0.34)
  Overall unpleasantness | 2.98 (0.34) | 3.55 (0.35)
  Intense deep pain | 3.33 (0.37) | 3.77 (0.37)
  Intense surface pain | 1.61 (0.28) | 1.82 (0.29)
  Average surface pain | 0.99 (0.15) | 1.05 (0.15)
  Average deep pain | 2.38 (0.29) | 2.55 (0.29)
  Average paroxysmal pain | 1.78 (0.25) | 2.06 (0.25)
Statistical Analysis 1: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; Intense: the difference between Lidoderm and placebo was compared by combining data for patients receiving the respective treatment regardless of the randomized study sequence. The endpoint was analyzed by linear mixed effects models incorporating treatment, period, sequence, and first-order carryover as fixed effects, and patient nested within sequence as a random effect. P-value for the random effect (s2) is from the Wald Z-test for the covariance parameter estimates; Test type: Superiority or Other; p = 0.4498, Linear mixed effects model — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = -0.22, 95% CI [-0.80 to 0.36] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; Sharp: the difference between Lidoderm and placebo was compared by combining data for patients receiving the respective treatment regardless of the randomized study sequence. The endpoint was analyzed by linear mixed effects models incorporating treatment, period, sequence, and first-order carryover as fixed effects, and patient nested within sequence as a random effect. P-value for the random effect (s2) is from the Wald Z-test for the covariance parameter estimates; Test type: Superiority or Other; p = 0.1065, Linear mixed effect models — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = -0.50, 95% CI [-1.11 to 0.11] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Lidoderm (Lidocaine 5% Patch); Hot: the difference between Lidoderm and placebo was compared by combining data for patients receiving the respective treatment regardless of the randomized study sequence. The endpoint was analyzed by linear mixed effects models incorporating treatment, period, sequence, and first-order carryover as fixed effects, and patient nested within sequence as a random effect. P-value for the random effect (s2) is from the Wald Z-test for the covariance parameter estimates; Test type: Superiority or Other; p = 0.0484, Linear mixed effects models — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = -0.47, 95% CI [-0.94 to -0.00] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Lidoderm (Lidocaine 5% Patch); Dull: the difference between Lidoderm and placebo was compared by combining data for patients receiving the respective treatment regardless of the randomized study sequence. The endpoint was analyzed by linear mixed effects models incorporating treatment, period, sequence, and first-order carryover as fixed effects, and patient nested within sequence as a random effect. P-value for the random effect (s2) is from the Wald Z-test for the covariance parameter estimates; Test type: Superiority or Other; p = 0.4973, Linear mixed effect models — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = -0.24, 95% CI [-0.93 to 0.46] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; Cold: the difference between Lidoderm and placebo was compared by combining data for patients receiving the respective treatment regardless of the randomized study sequence. The endpoint was analyzed by linear mixed effects models incorporating treatment, period, sequence, and first-order carryover as fixed effects, and patient nested within sequence as a random effect. P-value for the random effect (s2) is from the Wald Z-test for the covariance parameter estimates; Test type: Superiority or Other; p = 0.3966, Linear mixed effect models — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = 0.12, 95% CI [-0.16 to 0.41] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 6: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; Sensitive: the difference between Lidoderm and placebo was compared by combining data for patients receiving the respective treatment regardless of the randomized study sequence. The endpoint was analyzed by linear mixed effects models incorporating treatment, period, sequence, and first-order carryover as fixed effects, and patient nested within sequence as a random effect. P-value for the random effect (s2) is from the Wald Z-test for the covariance parameter estimates; Test type: Superiority or Other; p = 0.6941, Linear mixed effects model — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = -0.09, 95% CI [-0.53 to 0.35] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 7: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; Tender: the difference between Lidoderm and placebo was compared by combining data for patients receiving the respective treatment regardless of the randomized study sequence. The endpoint was analyzed by linear mixed effects models incorporating treatment, period, sequence, and first-order carryover as fixed effects, and patient nested within sequence as a random effect. P-value for the random effect (s2) is from the Wald Z-test for the covariance parameter estimates; Test type: Superiority or Other; p = 0.5664, Linear mixed effects models — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = 0.18, 95% CI [-0.45 to 0.82] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 8: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; Itchy: the difference between Lidoderm and placebo was compared by combining data for patients receiving the respective treatment regardless of the randomized study sequence. The endpoint was analyzed by linear mixed effects models incorporating treatment, period, sequence, and first-order carryover as fixed effects, and patient nested within sequence as a random effect. P-value for the random effect (s2) is from the Wald Z-test for the covariance parameter estimates; Test type: Superiority or Other; p = 0.6871, Linear mixed effects models — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = -0.09, 95% CI [-0.55 to 0.37] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 9: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; Shocking: the difference between Lidoderm and placebo was compared by combining data for patients receiving the respective treatment regardless of the randomized study sequence. The endpoint was analyzed by linear mixed effects models incorporating treatment, period, sequence, and first-order carryover as fixed effects, and patient nested within sequence as a random effect. P-value for the random effect (s2) is from the Wald Z-test for the covariance parameter estimates; Test type: Superiority or Other; p = 0.2318, Linear mixed effects models — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = -0.41, 95% CI [-1.08 to 0.27] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 10: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; Numb: the difference between Lidoderm and placebo was compared by combining data for patients receiving the respective treatment regardless of the randomized study sequence. The endpoint was analyzed by linear mixed effects models incorporating treatment, period, sequence, and first-order carryover as fixed effects, and patient nested within sequence as a random effect. P-value for the random effect (s2) is from the Wald Z-test for the covariance parameter estimates; Test type: Superiority or Other; p = 0.3383, Linear mixed effects models — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = -0.21, 95% CI [-0.64 to 0.22] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 11: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; Electrical: the difference between Lidoderm and placebo was compared by combining data for patients receiving the respective treatment regardless of the randomized study sequence. The endpoint was analyzed by linear mixed effects models incorporating treatment, period, sequence, and first-order carryover as fixed effects, and patient nested within sequence as a random effect. P-value for the random effect (s2) is from the Wald Z-test for the covariance parameter estimates; Test type: Superiority or Other; p = 0.8740, Linear mixed effects models — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = 0.05, 95% CI [-0.63 to 0.73] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 12: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; Tingling: the difference between Lidoderm and placebo was compared by combining data for patients receiving the respective treatment regardless of the randomized study sequence. The endpoint was analyzed by linear mixed effects models incorporating treatment, period, sequence, and first-order carryover as fixed effects, and patient nested within sequence as a random effect. P-value for the random effect (s2) is from the Wald Z-test for the covariance parameter estimates; Test type: Superiority or Other; p = 0.9990, Linear mixed effects models — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = -0.00, 95% CI [-0.54 to 0.54] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 13: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; Cramping: the difference between Lidoderm and placebo was compared by combining data for patients receiving the respective treatment regardless of the randomized study sequence. The endpoint was analyzed by linear mixed effects models incorporating treatment, period, sequence, and first-order carryover as fixed effects, and patient nested within sequence as a random effect. P-value for the random effect (s2) is from the Wald Z-test for the covariance parameter estimates; Test type: Superiority or Other; p = 0.4183, Linear mixed effects models — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = -0.25, 95% CI [-0.85 to 0.36] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 14: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; Radiating: the difference between Lidoderm and placebo was compared by combining data for patients receiving the respective treatment regardless of the randomized study sequence. The endpoint was analyzed by linear mixed effects models incorporating treatment, period, sequence, and first-order carryover as fixed effects, and patient nested within sequence as a random effect. P-value for the random effect (s2) is from the Wald Z-test for the covariance parameter estimates; Test type: Superiority or Other; p = 0.8227, Linear mixed effects models — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = -0.07, 95% CI [-0.71 to 0.57] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 15: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; Throbbing: the difference between Lidoderm and placebo was compared by combining data for patients receiving the respective treatment regardless of the randomized study sequence. The endpoint was analyzed by linear mixed effects models incorporating treatment, period, sequence, and first-order carryover as fixed effects, and patient nested within sequence as a random effect. P-value for the random effect (s2) is from the Wald Z-test for the covariance parameter estimates; Test type: Superiority or Other; p = 0.5870, Linear mixed effects models — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = 0.18, 95% CI [-0.48 to 0.85] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 16: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; Aching: the difference between Lidoderm and placebo was compared by combining data for patients receiving the respective treatment regardless of the randomized study sequence. The endpoint was analyzed by linear mixed effects models incorporating treatment, period, sequence, and first-order carryover as fixed effects, and patient nested within sequence as a random effect. P-value for the random effect (s2) is from the Wald Z-test for the covariance parameter estimates; Test type: Superiority or Other; p = 0.2181, Linear mixed effects models — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = -0.44, 95% CI [-1.15 to 0.27] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 17: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; Heavy: the difference between Lidoderm and placebo was compared by combining data for patients receiving the respective treatment regardless of the randomized study sequence. The endpoint was analyzed by linear mixed effects models incorporating treatment, period, sequence, and first-order carryover as fixed effects, and patient nested within sequence as a random effect. P-value for the random effect (s2) is from the Wald Z-test for the covariance parameter estimates; Test type: Superiority or Other; p = 0.6276, Linear mixed effects models — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = -0.13, 95% CI [-0.68 to 0.42] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 18: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; Overall unpleasantness: the difference between Lidoderm and placebo was compared by combining data for patients receiving the respective treatment regardless of the randomized study sequence. The endpoint was analyzed by linear mixed effects models incorporating treatment, period, sequence, and first-order carryover as fixed effects, and patient nested within sequence as a random effect. P-value for the random effect (s2) is from the Wald Z-test for the covariance parameter estimates; Test type: Superiority or Other; p = 0.0917, Linear mixed effects models — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = -0.57, 95% CI [-1.23 to 0.09] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 19: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; Intense deep pain: the difference between Lidoderm and placebo was compared by combining data for patients receiving the respective treatment regardless of the randomized study sequence. The endpoint was analyzed by linear mixed effects models incorporating treatment, period, sequence, and first-order carryover as fixed effects, and patient nested within sequence as a random effect. P-value for the random effect (s2) is from the Wald Z-test for the covariance parameter estimates; Test type: Superiority or Other; p = 0.2089, Linear mixed effects models — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = -0.44, 95% CI [-1.13 to 0.25] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 20: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; Intense surface pain: the difference between Lidoderm and placebo was compared by combining data for patients receiving the respective treatment regardless of the randomized study sequence. The endpoint was analyzed by linear mixed effects models incorporating treatment, period, sequence, and first-order carryover as fixed effects, and patient nested within sequence as a random effect. P-value for the random effect (s2) is from the Wald Z-test for the covariance parameter estimates; Test type: Superiority or Other; p = 0.4188, Linear mixed effects models — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = -0.22, 95% CI [-0.75 to 0.31] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 21: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; Average surface pain: the difference between Lidoderm and placebo was compared by combining data for patients receiving the respective treatment regardless of the randomized study sequence. The endpoint was analyzed by linear mixed effects models incorporating treatment, period, sequence, and first-order carryover as fixed effects, and patient nested within sequence as a random effect. P-value for the random effect (s2) is from the Wald Z-test for the covariance parameter estimates; Test type: Superiority or Other; p = 0.6959, Linear mixed effects models — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = -0.05, 95% CI [-0.32 to 0.21] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 22: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; Average deep pain: the difference between Lidoderm and placebo was compared by combining data for patients receiving the respective treatment regardless of the randomized study sequence. The endpoint was analyzed by linear mixed effects models incorporating treatment, period, sequence, and first-order carryover as fixed effects, and patient nested within sequence as a random effect. P-value for the random effect (s2) is from the Wald Z-test for the covariance parameter estimates; Test type: Superiority or Other; p = 0.4806, Linear mixed effects models — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = -0.17, 95% CI [-0.64 to 0.30] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 23: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; Average paroxysmal pain: the difference between Lidoderm and placebo was compared by combining data for patients receiving the respective treatment regardless of the randomized study sequence. The endpoint was analyzed by linear mixed effects models incorporating treatment, period, sequence, and first-order carryover as fixed effects, and patient nested within sequence as a random effect. P-value for the random effect (s2) is from the Wald Z-test for the covariance parameter estimates; Test type: Superiority or Other; p = 0.2291, Linear mixed effects models — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = -0.28, 95% CI [-0.74 to 0.18] — [estimate comment as in outcome 4, analysis 1]

7. Secondary Outcome: Patient Global Impression of Change From Baseline in Osteoarthritis (OA) Pain
Description: Patients rated their overall impression of change from Baseline to the end of each period during the double-blind treatment period, including premature discontinuation. Change was rated using a categorical scale indicating: "very much worse" (0); "much worse" (1); "minimally worse" (2); "no change" (3); "minimally improved" (4); "much improved" (5); and "very much improved" (6).
Time Frame: Baseline, Period 1 (up to 4 weeks), Period 2 (up to 4 weeks), Period 3 (up to 4 weeks)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Sequence: Lidoderm - Placebo - Placebo (LPP) | Sequence: Placebo - Lidoderm - Lidoderm (PLL)
Number analyzed (Participants) | 21 | 21
Participants
  6-Very Much Impr, Period 1 (LPP, N=21; PLL, N=21) | 3 | 5
  6-Very Much Impr., Period 2 (LPP, N=19; PLL, N=20) | 3 | 2
  6-Very Much Impr., Period 3 (LPP, N=19; PLL, N=19) | 4 | 4
  5-Much Improved, Period 1 (LPP, N=21; PLL, N=21) | 6 | 8
  5-Much Improved, Period 2 (LPP, N=19; PLL, N=20) | 9 | 8
  5-Much Improved, Period 3 (LPP, N=19; PLL, N=19) | 8 | 10
  4-Mini. Improved, Period 1 (LPP, N=21; PLL, N=21) | 7 | 4
  4-Mini. Improved, Period 2 (LPP, N=19; PLL, N=20) | 3 | 6
  4-Mini. Improved, Period 3 (LPP, N=19; PLL, N=19) | 3 | 3
  3-No Change, Period 1 (LPP, N=21; PLL, N=21) | 5 | 1
  3-No Change, Period 2 (LPP, N=19; PLL, N=20) | 1 | 2
  3-No Change, Period 3 (LPP, N=19; PLL, N=19) | 4 | 2
  2-Minimally Worse, Period 1 (LPP, N=21; PLL,N=19) | 0 | 3
  2-Minimally Worse, Period 2 (LPP, N=19; PLL, N=20) | 1 | 1
  2-Minimally Worse, Period 3 (LPP, N=19; PLL, N=19) | 0 | 0
  1-Much Worse, Period 1 (LPP, N=21; PLL, N=21) | 0 | 0
  1-Much Worse, Period 2 (LPP, N=19; PLL, N=20) | 2 | 0
  1-Much Worse, Period 3 (LPP, N=19; PLL, N=19) | 0 | 0
  0-Very Much Worse, Period 1 (LPP,N=21; PLL, N=21) | 0 | 0
  0-Very Much Worse, Period 2 (LPP, N=19; PLL, N=20) | 0 | 1
  0-Very Much Worse, Period 3 (LPP, N=19; PLL, N=19) | 0 | 0
Statistical Analysis 1: Comparison: Sequence: Lidoderm - Placebo - Placebo (LPP) vs Sequence: Placebo - Lidoderm - Lidoderm (PLL); Global impression of change from baseline with the lidocaine patch 5% and placebo patch were compared by combining data for patients receiving the respective treatment regardless of the randomized study sequence. An ordinal multinomial regression model was performed with sequence, period, treatment, carry over effect as fixed effects, with repeated measures taken on patient within sequence; Test type: Superiority or Other; p = 0.3185, Regression, Linear — All statistical tests were 2-sided with a significance level of alpha=0.05; Odds Ratio (OR) = 1.32, 95% CI [0.77 to 2.27] — The Odds Ratio (OR) provided is the ratio of Lidoderm to Placebo

8. Secondary Outcome: Investigator Global Impression of Change From Baseline in Osteoarthritis (OA) Pain
Description: Investigators rated their overall impression of change from Baseline to the end of each period during the double-blind treatment period, including premature discontinuation. Change was rated using a categorical scale ranging from "very much worse" to "very much improved." A similar questionnaire was completed by the Investigator.
Time Frame: Baseline, Period 1 (up to 4 weeks), Period 2 (up to 4 weeks), Period 3 (up to 4 weeks)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Sequence: Lidoderm - Placebo - Placebo (LPP) | Sequence: Placebo - Lidoderm - Lidoderm (PLL)
Number analyzed (Participants) | 21 | 21
Participants
  6-Very Much Impr, Period 1 (LPP, N=21; PLL, N=21) | 3 | 4
  6-Very Much Impr, Period 2 (LPP, N=19; PLL, N=20) | 2 | 3
  6-Very Much Impr, Period 3 (LPP, N=19; PLL, N=19) | 5 | 4
  5-Much Improved, Period 1 (LPP, N=21; PLL, N=21) | 7 | 9
  5-Much Improved, Period 2 (LPP, N=19; PLL, N=20) | 10 | 8
  5-Much Improved, Period 3 (LPP, N=19; PLL, N=19) | 7 | 8
  4-Min. Improved, Period 1 (LPP, N=21; PLL, N=21) | 4 | 2
  4-Min. Improved, Period 2 (LPP, N=19; PLL, N=20) | 3 | 7
  4-Min. Improved, Period 3 (LPP, N=19; PLL, N=19) | 4 | 4
  3-No Change, Period 1 (LPP, N=21; PLL, N=21) | 3 | 2
  3-No Change, Period 2 LPP, N=19; PLL, N=20) | 0 | 1
  3-No Change, Period 3 (LPP, N=19; PLL, N=19) | 1 | 2
  2-Minimally Worse, Period 1 (LPP, N=21; PLL, N=21) | 3 | 3
  2-Minimally Worse, Period 2 (LPP, N=19; PLL, N=20) | 1 | 0
  2-Minimally Worse, Period 3 (LPP, N=19; PLL, N=19) | 0 | 1
  1-Much Worse, Period 1 (LPP, N=21; PLL, N=21) | 1 | 1
  1-Much Worse, Period 2 (LPP, N=19; PLL, N=20) | 3 | 0
  1-Much Worse, Period 3 (LPP, N=19; PLL, N=19) | 1 | 0
  0-Very Much Worse, Period 1 (LPP, N=21; PLL, N=21) | 0 | 0
  0-Very Much Worse, Period 2 (LPP, N=19; PLL, N=20) | 0 | 1
  0-Very Much Worse, Period 3 (LPP, N=19; PLL, N=19) | 1 | 0
Statistical Analysis 1: Comparison: Sequence: Lidoderm - Placebo - Placebo (LPP) vs Sequence: Placebo - Lidoderm - Lidoderm (PLL); [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.4748, Regression, Linear — All statistical tests were 2-sided with a significance level of alpha=0.05; Odds Ratio (OR) = 1.22, 95% CI [0.72 to 2.06] — The odds ratio (OR) provided is the ratio of Lidoderm to Placebo

9. Other Pre Specified Outcome: Overall Treatment Difference in LSMeans of Beck Depression Inventory Second Edition (BDI-II) Total Score
Description: The BDI-II is a 21-item self-report instrument intended to assess the existence and severity of symptoms of depression. Patients were to consider each item as it related to the way they felt for the previous 2 weeks. Each of the 21 items corresponding to a symptom of depression was summed to give a single score for the BDI-II, with a 4-point scale for each item ranging from 0-3. A total score of 0-13 is minimal, 14-19 is mild, 20-28 is moderate, and 29-63 is severe. Values were based on measurements taken at Screening, at Baseline (Visit 3), and at the end of each period.
Time Frame: Baseline and end of treatment period (up to 4 weeks)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Lidoderm (Lidocaine 5% Patch) | Placebo Patch
Number analyzed (Participants) | 21 | 21
Units on a scale | 4.41 (0.39) | 4.29 (0.39)
Statistical Analysis 1: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; The overall treatment difference for the lidocaine patch 5% and placebo patch was compared by combining data for patients receiving the respective treatment regardless of randomized study sequence. The endpoint was analyzed by linear mixed effects models incorporating treatment, period, sequence, and first-order carryover as fixed effects, and patient nested within sequence as a random effect. P-value for the random effect (s2) is from the Wald Z-test for the covariance parameter estimates; Test type: Superiority or Other; p = 0.7839, Linear mixed effects models — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = 0.12, 95% CI [-0.74 to 0.98] — [estimate comment as in outcome 4, analysis 1]

10. Other Pre Specified Outcome: Quality of Life: Four Category Beck Depression Inventory Second Edition (BDI-II) Composite Score
Description: as for outcome 9
Time Frame: Screening, Baseline, Period 1 (up to 4 weeks), Period 2 (up to 4 weeks), Period 3 (up to 4 weeks)
Population: as for outcome 3
Measure: Number; unit: Participants
Groups:
- Sequence: Lidoderm - Placebo - Placebo (LPP): Lidoderm (lidocaine 5% patch) 10cm X 14cm patches each on the front and back of the index knee every 24 hours (q24h) for 4 weeks followed by matching placebo 10cm x 14cm patches each on the front and back of the index knee q24h for up to 8 weeks
Arm/Group | Sequence: Lidoderm - Placebo - Placebo (LPP) | Sequence: Placebo - Lidoderm - Lidoderm (PLL)
Number analyzed (Participants) | 21 | 21
Participants
  Minimal at Screening (LPP, N=21; PLL, N=21) | 21 | 20
  Minimal at Baseline (LPP, N=21; PLL, N=21) | 21 | 20
  Minimal, end of Period 1 (LPP, N=21; PLL, N=21) | 21 | 19
  Minimal, end of Period 2 (LPP, N=19; PLL, N=20) | 19 | 20
  Minimal, end of Period 3 (LPP, N=19; PLL, N=19) | 19 | 19
  Mild at Screening (LPP, N=21; PLL, N=21) | 0 | 1
  Mild at Baseline (LPP, N=21; PLL, N=21) | 0 | 1
  Mild, end of Period 1 (LPP, N=21; PLL, N=21) | 0 | 1
  Mild, end of Period 2 (LPP, N=19; PLL, N=20) | 0 | 0
  Mild, end of Period 3 (LPP, N=19; PLL, N=19) | 0 | 0
  Moderate at Screening (LPP, N=21; PLL, N=21) | 0 | 0
  Moderate at Baseline (LPP, N=21; PLL, N=21) | 0 | 0
  Moderate, end of Period 1 (LPP, N=21; PLL, N=21) | 0 | 1
  Moderate, end of Period 2 (LPP, N=19; PLL, N=20) | 0 | 0
  Moderate, end of Period 3 (LPP, N=19; PLL, N=19) | 0 | 0
  Severe at Screening (LPP, N=21; PLL, N=21) | 0 | 0
  Severe at Baseline (LPP, N=21; PLL, N=21) | 0 | 0
  Severe, end of Period 1 (LPP, N=21; PLL, N=21) | 0 | 0
  Severe, end of Period 2 (LPP, N=19; PLL, N=20) | 0 | 0
  Severe, end of Period 3 (LPP, N=19; PLL, N=19) | 0 | 0

11. Other Pre Specified Outcome: Overall Treatment Difference in LSMeans for Continuous EuroQol Quality of Life Instrument (EQ-5D) Index Scores
Description: Health status was assessed using the EuroQol Quality of Life Instrument (EQ-5D). Patients completed the EQ-5D assessment at Baseline (Day 0) and at each clinic visit (at least every 4 weeks) or at premature discontinuation. Values of the EQ-5D index score range from -1 (worst) to 1 (best).
Time Frame: Baseline, Period 1 (up to 4 weeks), Period 2 (up to 4 weeks), Period 3 (up to 4 weeks), or Premature Discontinuation
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Lidoderm (Lidocaine 5% Patch) | Placebo Patch
Number analyzed (Participants) | 21 | 21
Units on a scale | 0.82 (0.01) | 0.81 (0.01)
Statistical Analysis 1: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.3773, Linear mixed effects model — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = 0.01, 95% CI [-0.02 to 0.04] — [estimate comment as in outcome 4, analysis 1]

12. Secondary Outcome: Patient Global Assessment of Treatment Satisfaction
Description: At the end of each period, patients rated their overall satisfaction with study treatment using a 5-point categorical scale indicating: 0 - very dissatisfied; 1 - dissatisfied; 2 - no preference; 3 - satisfied; and 4 - very satisfied.
Time Frame: Baseline, Period 1 (up to 4 weeks), Period 2 (up to 4 weeks), Period 3 (up to 4 weeks)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Sequence: Lidoderm - Placebo - Placebo (LPP) | Sequence: Placebo - Lidoderm - Lidoderm (PLL)
Number analyzed (Participants) | 21 | 21
Participants
  4-Very Satisfied, Period 1 (LPP, N=21; PLL, N=21) | 12 | 9
  4-Very Satisfied, Period 2 (LPP, N=19; PLL, N=20) | 8 | 10
  4-Very Satisfied, Period 3 (LPP, N=19; PLL, N=20) | 12 | 12
  3-Satisfied, Period 1 (LPP, N=21; PLL, N=21) | 7 | 8
  3-Satisfied, Period 2 (LPP, N=19; PLL, N=20) | 9 | 6
  3-Satisfied, Period 3 (LPP, N=19; PLL, N=20) | 5 | 6
  2-No Preference, Period 1 (LPP, N=21; PLL, N=21) | 1 | 3
  2-No Preference, Period 2 (LPP, N=19; PLL, N=20) | 0 | 3
  2-No Preference, Period 3 (LPP, N=19; PLL, N=20) | 1 | 1
  1-Dissatisfied, Period 1 (LPP, N=21; PLL, N=21) | 1 | 1
  1-Dissatisfied, Period 2 (LPP, N=19; PLL, N=20) | 2 | 0
  1-Dissatisfied, Period 3 (LPP, N=19; PLL, N=20) | 0 | 0
  0-Very Dissatisfied, Per. 1 (LPP, N=21; PLL, N=21) | 0 | 0
  0-Very Dissatisfied, Per. 2 (LPP, N=19; PLL, N=20) | 0 | 1
  0-Very Dissatisfied, Per. 3 (LPP, N=19; PLL, N=19) | 1 | 0
Statistical Analysis 1: Comparison: Sequence: Lidoderm - Placebo - Placebo (LPP) vs Sequence: Placebo - Lidoderm - Lidoderm (PLL); Treatment satisfaction with the lidocaine patch 5% and placebo patch were compared by combining data for patients receiving the respective treatment regardless of the randomized study sequence. An ordinal multinomial regression model was performed with sequence, period, treatment, carry over effect as fixed effects, with repeated measures taken on patient within sequence; Test type: Superiority or Other; p = 0.2605, Regression, Linear — All statistical tests were 2-sided with a significance level of alpha=0.05; Odds Ratio (OR) = 0.71, 95% CI [0.38 to 1.30] — The odds ratio (OR) provided is the ratio of Lidoderm to Placebo

13. Secondary Outcome: Investigator Global Assessment of Treatment Satisfaction
Description: At the end of each period, investigators rated their overall satisfaction with study treatment using a 5-point categorical scale ranging from 0 (very dissatisfied) to 4 (very satisfied).
Time Frame: Baseline, Period 1 (up to 4 weeks), Period 2 (up to 4 weeks), Period 3 (up to 4 weeks)
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Sequence: Lidoderm - Placebo - Placebo (LPP) | Sequence: Placebo - Lidoderm - Lidoderm (PLL)
Number analyzed (Participants) | 21 | 21
Participants
  4-Very Satisfied, Period 1 (LPP, N=21; PLL,N=21) | 7 | 6
  4-Very Satisfied, Period 2 (LPP, N=19; PLL, N=20) | 5 | 8
  4-Very Satisfied, Period 3 (LPP, N=19; PLL, N=19) | 8 | 11
  3-Satisfied, Period 1 (LPP, N=21; PLL,N=21) | 8 | 9
  3-Satisfied, Period 2 (LPP, N=19; PLL, N=20) | 11 | 10
  3-Satisfied, Period 3 (LPP, N=19; PLL, N=19) | 9 | 5
  2-No Preference, Period 1 (LPP, N=21; PLL,N=21) | 1 | 1
  2-No Preference, Period 2 (LPP, N=19; PLL, N=20) | 1 | 1
  2-No Preference, Period 3 (LPP, N=19; PLL, N=19) | 1 | 2
  1-Dissatisfied, Period 1 (LPP, N=21; PLL,N=21) | 4 | 5
  1-Dissatisfied, Period 2 (LPP, N=19; PLL, N=20) | 2 | 0
  1-Dissatisfied, Period 3 (LPP, N=19; PLL, N=19) | 0 | 1
  0-Very Dissatisfied, Period 1 (LPP,N=21; PLL,N=21) | 1 | 0
  0-Very Dissatisfied, Period 2 (LPP,N=19; PLL,N=20) | 0 | 1
  0-Very Dissatisfied, Period 3 (LPP,N=19; PLL,N=19) | 1 | 0
Statistical Analysis 1: Comparison: Sequence: Lidoderm - Placebo - Placebo (LPP) vs Sequence: Placebo - Lidoderm - Lidoderm (PLL); [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.3193, Regression, Linear — All statistical tests were 2-sided with a significance level of alpha=0.05; Odds Ratio (OR) = 0.76, 95% CI [0.44 to 1.30] — The odds ratio (OR) provided is the ratio of Lidoderm to Placebo

14. Other Pre Specified Outcome: Overall Treatment Difference in LSMeans for Continuous EuroQol Quality of Life Instrument (EQ-5D) Health Status Today Using a Visual Analog Scale (VAS)
Description: Health status was assessed using the EuroQol Quality of Life Instrument (EQ-5D). Patients completed the EQ-5D assessment at Baseline and at the end of each period or at premature discontinuation. Values of the continuous EQ-5D health state today (VAS) ranged from 0 (worst imaginable health state) to 100 (best imaginable health state).
Time Frame: Baseline, Period 1 (up to 4 weeks), Period 2 (up to 4 weeks), Period 3 (up to 4 weeks), or Premature Discontinuation
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Lidoderm (Lidocaine 5% Patch) | Placebo Patch
Number analyzed (Participants) | 21 | 21
Units on a scale | 81.1 (1.25) | 79.4 (1.26)
Statistical Analysis 1: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.1378, Linear mixed effects model — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = 1.74, 95% CI [-0.57 to 4.04] — [estimate comment as in outcome 4, analysis 1]

15. Other Pre Specified Outcome: Quality of Life: Three-Category EuroQol Quality of Life Instrument (EQ-5D) General Health Today Compared to Last 12 Months
Description: Health status was assessed using the EuroQol Quality of Life Instrument (EQ-5D). Patients completed the EQ-5D assessment at Baseline and at the end of each period or at premature discontinuation. Categories included Better, Much the Same, and Worse.
Time Frame: Baseline, Period 1 (up to 4 weeks), Period 2 (up to 4 weeks), Period 3 (up to 4 weeks), or Premature Discontinuation
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Sequence: Lidoderm - Placebo - Placebo (LPP) | Sequence: Placebo - Lidoderm - Lidoderm (PLL)
Number analyzed (Participants) | 21 | 21
Participants
  Better Baseline (LPP, N=21; PLL, N=21) | 11 | 4
  Better Period 1 (LPP, N=21; PLL, N=21) | 7 | 5
  Better Period 2 (LPP, N=19; PLL, N=20) | 8 | 4
  Better Period 3 (LPP, N=19; PLL, N=19) | 9 | 6
  Much the Same Baseline (LPP, N=21; PLL, N=21) | 10 | 17
  Much the Same Period 1 (LPP, N=21; PLL, N=21) | 14 | 15
  Much the Same Period 2 (LPP, N=19; PLL, N=20) | 10 | 16
  Much the Same Period 3 (LPP, N=19; PLL, N=19) | 9 | 12
  Worse Baseline (LPP, N=21; PLL, N=21) | 0 | 0
  Worse Period 1 (LPP, N=21; PLL, N=21) | 0 | 1
  Worse Period 2 (LPP, N=19; PLL, N=20) | 1 | 0
  Worse Period 3 (LPP, N=19; PLL, N=19) | 0 | 1
Statistical Analysis 1: Comparison: Sequence: Lidoderm - Placebo - Placebo (LPP) vs Sequence: Placebo - Lidoderm - Lidoderm (PLL); Test type: Superiority or Other; p = 0.6833, Regression, Logistic — All statistical tests were 2-sided with a significance level of alpha=0.05; An ordinal multinomial regression model was performed with sequence, period, treatment, carry over effect as fixed effects; Odds Ratio (OR) = 0.88, 95% CI [0.47 to 1.65] — The Odds Ratio (OR) provided is the ratio of Lidoderm to Placebo

16. Other Pre Specified Outcome: Overall Treatment Difference in LSMeans for Verran Snyder-Halpern (VSH) Sleep Scale
Description: The VSH Sleep Scale is contained in a 15 item self-report instrument that measures the quality of a patient's sleep over the last 24 hours. Each item is scored on a 0-100 visual analog scale. The VSH is categorized into 3 sleep scales: disturbance (which measures delays and interruptions in sleep)[maximum score = 700], effectiveness (which measures how well sleep refreshed the individual) [maximum score = 600], and supplementation (which measures the need for napping) [maximum score = 400]. The higher the score the greater the value of the sleep characteristic for that patient.
Time Frame: Baseline, Period 1 (up to 4 weeks), Period 2 (up to 4 weeks), Period 3 (up to 4 weeks)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Lidoderm (Lidocaine 5% Patch) | Placebo Patch
Number analyzed (Participants) | 21 | 21
Units on a scale
  Disturbance | 246 (13.7) | 224 (13.9)
  Effectiveness | 303 (9.69) | 302 (9.85)
  Supplementation | 49.7 (7.62) | 41.4 (7.76)
Statistical Analysis 1: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; Disturbance: the overall treatment difference for Lidoderm and placebo patch was compared by combining data for patients receiving the respective treatment regardless of randomized study sequence. The endpoint was analyzed by linear mixed effects models incorporating treatment, period, sequence, and first-order carryover as fixed effects, and patient nested within sequence as a random effect. P-value for the random effect (s2) is from the Wald Z-test for the covariance parameter estimates; Test type: Superiority or Other; p = 0.1143, Linear mixed effects models — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = 22.16, 95% CI [-5.48 to 49.8] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 2: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; Effectiveness: the overall treatment difference for Lidoderm and placebo patch was compared by combining data for patients receiving the respective treatment regardless of randomized study sequence. The endpoint was analyzed by linear mixed effects models incorporating treatment, period, sequence, and first-order carryover as fixed effects, and patient nested within sequence as a random effect. P-value for the random effect (s2) is from the Wald Z-test for the covariance parameter estimates; Test type: Superiority or Other; p = 0.9108, Linear mixed effects models — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = 1.18, 95% CI [-19.8 to 22.2] — [estimate comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Lidoderm (Lidocaine 5% Patch) vs Placebo Patch; Supplementation: the overall treatment difference for Lidoderm and placebo patch was compared by combining data for patients receiving the respective treatment regardless of randomized study sequence. The endpoint was analyzed by linear mixed effects models incorporating treatment, period, sequence, and first-order carryover as fixed effects, and patient nested within sequence as a random effect. P-value for the random effect (s2) is from the Wald Z-test for the covariance parameter estimates; Test type: Superiority or Other; p = 0.3769, Linear mixed effects models — All statistical tests were 2-sided with a significance level of alpha=0.05; Mean Difference (Net) = 8.31, 95% CI [-10.3 to 27.0] — [estimate comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) were recorded from the beginning of the active Run-in Period through 30 days post-study completion/early termination; a period lasting up to 20 weeks in total.
Description: The safety population included all patients who received study medication during the study and did not return all study medication unopened.
Groups:
- Run-In Period With Lidoderm (Lidocaine 5% Patch): Treatment-Emergent Adverse Events (TEAEs) reported by subjects on Lidoderm (lidocaine 5% patch) during the active treatment Run-in Period.
  A treatment-emergent AE (TEAE) is any condition that was not present prior to treatment with study medication, but appeared following treatment, was present at treatment initiation, but worsened during treatment, or was present at treatment initiation, but resolved and then reappeared while the individual was on treatment (regardless of the intensity of the AE when the treatment was initiated).
- Double-Blind Treatment Period With Lidoderm: Treatment-Emergent Adverse Events (TEAEs) reported by subjects on Lidoderm (lidocaine 5% patch) during the Double-blind Treatment Period.
  A treatment-emergent AE (TEAE) is any condition that was not present prior to treatment with study medication, but appeared following treatment, was present at treatment initiation, but worsened during treatment, or was present at treatment initiation, but resolved and then reappeared while the individual was on treatment (regardless of the intensity of the AE when the treatment was initiated).
  *NOTE: two subjects randomized to the treatment sequence Placebo - Lidoderm - Lidoderm (PLL) discontinued from the study during treatment with Placebo (Period 1); therefore, the number of subjects included in the safety analysis by treatment group (Lidoderm) is equal to 91.
- Double-Blind Active Treatment Period With Placebo: Treatment-Emergent Adverse Events (TEAEs) reported by subjects on Placebo during the Double-blind Treatment Period.
  A treatment-emergent AE (TEAE) is any condition that was not present prior to treatment with study medication, but appeared following treatment, was present at treatment initiation, but worsened during treatment, or was present at treatment initiation, but resolved and then reappeared while the individual was on treatment (regardless of the intensity of the AE when the treatment was initiated).
  **NOTE: two subjects randomized to the treatment sequence Lidoderm - Placebo - Placebo (PLL) discontinued from the study during treatment with Lidoderm (Period 1); therefore, the number of subjects included in the safety analysis by treatment group (Placebo) is equal to 91.
Arm/Group | Run-In Period With Lidoderm (Lidocaine 5% Patch) | Double-Blind Treatment Period With Lidoderm | Double-Blind Active Treatment Period With Placebo
Serious Adverse Events (participants affected / at risk) | 1/169 | 1/91 | 1/91
Other Adverse Events (participants affected / at risk) | 51/169 | 24/91 | 23/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-In Period With Lidoderm (Lidocaine 5% Patch) (N=169) | Double-Blind Treatment Period With Lidoderm (N=91) | Double-Blind Active Treatment Period With Placebo (N=91)
Pneumonia (Infections and infestations) | 1 | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Run-In Period With Lidoderm (Lidocaine 5% Patch) (N=169) | Double-Blind Treatment Period With Lidoderm (N=91) | Double-Blind Active Treatment Period With Placebo (N=91)
Application site dermatitis (General disorders) | 2 | 0 | 0
Application site erythema (General disorders) | 2 | 1 | 2
Oedema peripheral (General disorders) | 2 | 1 | 0
Pain (General disorders) | 2 | 0 | 0
Pyrexia (General disorders) | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 2 | 3
Sinusitis (Infections and infestations) | 2 | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Headache (Nervous system disorders) | 3 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0
Application site reaction (General disorders) | 1 | 4 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1 | 1
Ear infection (Infections and infestations) | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 1
Keratitis herpetic (Infections and infestations) | 0 | 0 | 1
Otitis media (Infections and infestations) | 0 | 0 | 1
Vaginal candidiasis (Infections and infestations) | 0 | 0 | 1
Application site oedema (General disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 1
Renal cyst (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 1
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 1 | 0
Application site swelling (General disorders) | 1 | 0 | 0
Application site vesicles (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Stomach discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Nail pigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Burning sensation (Nervous system disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Burns first degree (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0
Anger (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Peripheral coldness (Vascular disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to operational issues, the modified intent-to-treat (MITT) population, consisting of all intent-to-treat (ITT) patients randomized on or after January 22, 2008, was added to the analysis plan; all efficacy data are presented for this population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Delay of 12-18 months from Completion Date to publish results from all sites, embargo of 60 to 180 days from the time communication is submitted to sponsor, and ability to redact confidential information (excluding results).